CLINICAL TRIAL: NCT04642794
Title: Management of Portoplenomesenteric Vein Thrombosis in Patients With Acute Pancreatitis : an Observational Study
Brief Title: Acute Pancreatitis and Thrombosis (PATHRO)
Acronym: PATHRO
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MR_PATHRO
Record Dates: First submitted 2020-11-17; First posted 2020-11-24 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Acute Necrotizing Pancreatitis; Portosplenomesenteric Venous Thrombosis
Keywords: acute necrotizing pancreatitis; acute pancreatitis; pancreas disease; anticoagulation; anticolagulant therapy; bleeding; Portosplenomesenteric Vein Thrombosis; splanchic venous thrombosis
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis; Pancreatic Diseases; Hemorrhage | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — patients admitted for AP with portosplenomesenteric vein thrombosis.

SUMMARY:
Severe acute pancreatitis (AP) is a pathology with high morbidity and mortality. Portosplenomesenteric vein thrombosis is a well-known local complication of AP with a variable incidence, which can reach up to 50% in case of severe AP. However, there is no specific recommendation regarding the management of Portosplenomesenteric vein thrombosis. By analogy to all venous thrombosis, the European Society of Gastroenterology recommends curative anticoagulation. However, the efficacy of curative anticoagulation has never been evaluated by prospective studies. In addition, bleeding complications during AP occur in approximately 10% of patients and are associated with a poor prognosis.

The investigators wish to conduct an observational multi-center study with epidemiologic aims, including all patients admitted for AP and with a diagnosis of portosplenomesenteric vein thrombosis. The aim of this study is to evaluate the therapeutic management of these patients, the efficacy and safety of anticoagulant treatment for the treatment of Portosplenomesenteric vein thrombosis, and their outcomes.

DETAILED DESCRIPTION:
The investigators will include prospectively all patients admitted for AP with a computed tomography diagnosis of portosplenomesenteric vein thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients (age > 18 years) with acute pancreatitis
* AND a diagnosis on CT injected with portal time of portosplenomesenteric vein thrombosis or laminated veins (without passage of blood flow through the vessel but without visible intraluminal thrombus) will be included.

Exclusion Criteria:

* Patient under guardianship
* Refusal to participate in research
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted for AP with portosplenomesenteric vein thrombosis
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
incidence of anticoagulation therapy | up to 12 months
  incidence defined as : the ratio of the number of patients on curative anticoagulant therapy to the number of patients admitted with AP and portosplenomesenteric vein thrombosis during the inclusion period

SECONDARY OUTCOMES:
evaluate the outcomes of Number of patients admitted for AP with portosplenomesenteric vein thrombosis | up to 12 months
hospital mortality at D28 | Day 28
  evaluate the hospitality mortality at D28 of patients admitted for AP with portosplenomesenteric vein
hospital mortality at D90 | Day 90
  evaluate the hospitality mortality at D90 of patients admitted for AP with portosplenomesenteric vein
hospital mortality at 6 months | 6 months
  evaluate the hospitality mortality at 6 months of patients admitted for AP with portosplenomesenteric vein
hospital mortality at 12 months | 12 months
  evaluate the hospitality mortality at 12 months of patients admitted for AP with portosplenomesenteric vein
incidence of portal cavernoma | up to 12 months
  evaluate the incidence of portal cavernoma of patients admitted for AP with portosplenomesenteric vein
incidence of type 2 diabetes secondary to AP | up to 12 months
  evaluate the incidence of type 2 diabetes secondary to AP of patients admitted for AP with portosplenomesenteric vein
incidence of occurrence of malabsorption | up to 12 months
  evaluate the incidence of occurrence of malabsorption of patients admitted for AP with portosplenomesenteric vein
incidence of digestive ischemia | up to 12 months
  evaluate the incidence of digestive ischemia of patients admitted for AP with portosplenomesenteric vein
incidence of hepatic ischemia | up to 12 months
  evaluate the incidence of hepatic ischemia of patients admitted for AP with portosplenomesenteric vein
incidence of pancreatic necrosis | up to 12 months
  evaluate the incidence of pancreatic necrosis of patients admitted for AP with portosplenomesenteric vein

CONTACTS AND LOCATIONS:
Overall Officials: GARRET Charlotte, MD, Principal Investigator — University hospital of Nantes
Locations (1):
- CHU de Nantes, Nantes, France